CLINICAL TRIAL: NCT00744744
Title: A CROSS-SECTIONAL STUDY OF PATIENT-REPORTED OUTCOMES FOR BLADDER CANCER PATIENTS WITH NON-INVASIVE DISEASE
Brief Title: Health-Related Quality of Life in Patients With Bladder Cancer
Status: Completed | Type: Observational
Sponsor: David Latini (Other)
Responsible Party: Sponsor-Investigator, David Latini, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: CDR0000600461; BCM-H-21350
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey
  Interventions: Other: informational intervention; Other: questionnaire administration; Procedure: management of therapy complications; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: informational intervention — Patient educational information
Other: questionnaire administration — Survey
Procedure: management of therapy complications — Survey
Procedure: psychosocial assessment and care — Survey
Procedure: quality-of-life assessment — Survey

SUMMARY:
RATIONALE: Gathering information about quality of life in patients with cancer may improve the ability to plan treatment and may help patients live more comfortably.

PURPOSE: This clinical trial is studying health-related quality of life in patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify aspects of survivorship experience that differ by clinical risk (low risk vs high risk) in patients with non-invasive bladder cancer.
* To collect and examine data on health-related quality of life (HRQOL) and symptom management.
* To analyze differences in outcomes between genders, stage and grade of disease, and recency of diagnosis (new diagnosis vs ≥ 6 month diagnosis).

OUTLINE: Patients undergo a 45-minute telephone interview to assess their current medical condition and psychological functioning (i.e., bladder cancer treatment history, levels of depression and anxiety, quality of life, self-efficacy, and perceived social support). Patients complete a series of questionnaires including the Lepore social constraint measure; REACH social support measure; self-report inventories assessing patient communication, relationship style, illness intrusiveness, fear of recurrence, and social constraint; Impact of Events scale; Brief Symptom Index-18 and Global Severity Index; EORTC QLQ-C30 (general health-related quality of life); and EORTC QLC-BLS24 (disease-specific health-related quality of life).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-invasive bladder cancer within the past 4 years

PATIENT CHARACTERISTICS:

* Not pregnant
* Able to read, speak, and understand English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons diagnosed with bladder cancer within 4 years of study entry
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Collection and examination of data on health-related quality of life and symptom management | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: David M. Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas, United States